CLINICAL TRIAL: NCT03892993
Title: Designing a Decision Aid to Help People With Medullary Thyroid Cancer Make Decisions With Their Doctors About Whether to Start or Stop New Drugs, Enroll in Clinical Trials, or Continue With Active Surveillance
Brief Title: Patient Decision Aid in Supporting Decision-Making About When to Start or Stop New Drugs, Join Clinical Trials, or Continue Active Surveillance in Patients With Medullary Thyroid Cancer and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0557; NCI-2019-00631 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0557 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-02-21; First posted 2019-03-27 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Gland Medullary Carcinoma
MeSH Terms: conditions — Carcinoma, Medullary | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (decision aid) (Experimental): Participants use decision aid and complete questionnaires.
  Interventions: Other: Decision Aid; Other: Questionnaire Administration

INTERVENTIONS:
Other: Decision Aid — Use decision aid
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial develops and studies how well a patient decision aid works in supporting decision-making about when to start or stop new drugs, join clinical trials, or continue active cancer monitoring for patients with medullary thyroid cancer and their caregivers. Developing a patient decision aid may help patients with medullary thyroid cancer make well-informed decisions about their cancer care and be able to discuss their preferences with their doctors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess patient/survivor, caregiver/family member, and provider decision-making needs.

II. To design and develop an initial patient decision aid prototype. III. To pilot test its acceptability. IV. To evaluate the acceptability and usability of the decision aid prototype from patients/survivors, caregivers and providers in a real world environment.

OUTLINE:

Participants use decision aid and complete questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or older
* Have or will face(d) this decision, including: Patient/survivor - who has medullary thyroid carcinoma, as determined by a clinician or documented in the Genetics of Endocrine Neoplasia Registry or sporadic (medullary thyroid carcinoma) MTC database; Caregiver/family member - of patient/survivor who has medullary thyroid carcinoma, as nominated by the patient/survivor; and Provider - who treats patients/survivors who have medullary thyroid carcinoma, as described above
* Able to speak, read, and write English
* Pregnant patients are included

Exclusion Criteria:

--Individuals with cognitive or psychological impairment (e.g., depression, anxiety, severe mental illness; as documented in the registry)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-04-09 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Needs assessment | Up to 1 year
  The research team will tabulate and summarize responses to the needs assessment questionnaire to identify priority design needs, and review open text areas for notable suggestions.
Decision aid design refining (storyboarding) | Up to 1 year
  During storyboarding, the research team will iteratively review the interviewers' notes regarding participant feedback, identify predominant recommendations for improvement, and make decisions to refine the decision aid design.
Decision aid acceptability | Up to 1 year post decision aid
  The research team will review the Think Aloud interview notes for potential opportunities for improvement. Responses to the post-decision aid acceptability questionnaire will be tabulated and summarized into tables for publication and presentation using Excel. The Stakeholder Advisory Panel will review responses to the post-decision aid acceptability questionnaire, to confirm that viewing the decision aid provides a balanced presentation of the options and is not likely to bias patients'/survivors' initial preferences.
Real World Evaluation | Up to 1 year post
  Responses to the participant characteristics will be tabulated and summarized for presentation and publication, as appropriate. The research team will tabulate and summarize responses to the needs assessment questionnaire to identify priority design needs and review open text areas for notable suggestions.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth G Grubbs, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org